CLINICAL TRIAL: NCT04374955
Title: The Effect of Probiotic Added to Maternal Diet on Infantile Colic and Intestinal Microbiota Content: A Randomized Controlled Trials
Brief Title: The Effect of Probiotic Added to Maternal Diet on Infantile Colic and Intestinal Microbiota Content
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Collaborators: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Aysu Yıldız Karaahmet, MsC, Halic University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: a6pu2f37
Record Dates: First submitted 2020-04-29; First posted 2020-05-05 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Infantile Colic; Microbial Colonization; Crying
Keywords: infantile colic, colic, probiotics, maternal diet, microbiota
MeSH Terms: conditions — Colic; Communicable Diseases; Crying

STUDY DESIGN:
Intervention Model Description: One blind, Randomized controlled Trials
Who Masked: Participant, Investigator
Masking Description: One-blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İnfantile colic (Experimental): Mothers of babies diagnosed with infantile colic in the intervention group will receive routine care and start taking probiotic products after the first stool of the babies and blood is taken for intestinal permeability and will continue for 15 days.
  Interventions: Dietary Supplement: Activia Probiotics Shot; Other: Routine care
- Control (Other): Mothers of babies diagnosed with infantile colic in the control group will receive routine care for 15 days after blood is taken for the first stool and intestinal permeability of the babies.
  Interventions: Other: Routine care

INTERVENTIONS:
Dietary Supplement: Activia Probiotics Shot — The product contains Actiregularis - at least 2x106 cfu / g.
  Arms: İnfantile colic
Other: Routine care — Routine care of the hospital will be provided.

SUMMARY:
This study aims to investigate the effect of probiotic added to the diet of mothers on infantile colic in the postpartum period and the content of the neonatal intestinal microbiota.

DETAILED DESCRIPTION:
Infantile colic, by definition, is defined as excessive crying in the afternoon or evening, with no specific reason, starting at the first weeks of newborn life, lasting at least 3 weeks, longer than 3 hours a day and more than 3 days a week. Infantile colic is a common newborn problem worldwide, affecting approximately 20% of infants. Although infantile colic is considered a self-limiting and benign problem, it is a stressful problem for both newborns and parents.

It is thought that the factors affecting infantile colic etiology may be the mode of delivery, diet, birth weight, intestinal contractions, lactose intolerance, food hypersensitivity, gas, parental misinterpretation of the normal crying model, or various combinations of the above. In recent years and related evidence, it has been suggested that motility disorder and intestinal neuronal hyperexcitability are the most important pathogenic factor in infantile colic etiology. However, increasing evidence suggests that changes in the gut microbiota may contribute to the development of this condition. By definition, microbiota is expressed as a collection of microorganisms within a certain environment or ecosystem. While the microbiota formation forms pathogenic, commensal and symbiotic microorganisms found in the human body, the formation of the intestinal microbiota (colonization with bacteria) begins in the womb, with the transition from the vagina at birth, this colonization continues intensely and the foundations of the intestinal microbiota are laid in the first 3 months of life. The ideal situation for the microbiota is that the beneficial and harmful bacteria in the intestinal flora stay in balance and form a healthy flora. While discussing what is a healthy microbiota, it is expressed as dysbiosis in case of beneficial and harmful flora in balance.

In infantile colic, when the microbial structure was evaluated, it was seen to be characterized by different microbial patterns. In the first 2 weeks of life, infants with infantile colic have been reported to have a lower variety and stability of the gut microbiota. When we look at the studies about microbiota, it was seen that especially in colic babies, E. coli bacteria is found to be excessive, and the amount of bifidobacterium and lactobacilli are decreased. In this case, coliforms are reported to cause pain by creating excessive gas and inflammatory lipopolysaccharides as a result of intestinal fermentation. In addition, studies show that babies with colic differ from those without babies without microbiota, whereas babies with colic showed low microbiota diversity and stability in the first weeks of life, and no difference was observed in the 3 to 4 month evaluations. Another important factor that plays a role in infantile colic etiology is diet. Breast milk, which is the most important food source for the newborn, has a unique and complex microbiological composition, rich oligosaccharide content, immunological factors and a probiotic (in the form of Bifidobacterium and Lactobacillus) and prebiotics that have the ability to ensure the content and mucosal development of the intestinal microbiota if taken in sufficient quantity. human milk oligosaccharide (HMO)) combination. When the microbial changes of the babies who were breastfed and fed formula formula were compared, it was observed that the rate of bifidobacterium and microorganism content of the babies who were breastfed were 10 times richer than the formula formula. In a study by Grönlund et al., 35-36 of pregnancy among 67 mothers. When the stool samples and breast milk samples taken from the baby during the first week and in the 1st month were evaluated, it was found that the content of bifidobacterium (the most dense bifidobacterium longum) in the stool content and milk of the mother was the most important factor affecting the type and amount of bifidobacterium in the baby's stool. These changes suggest that a condition of intestinal dysbiosis may play a role in the expression of infantile colic symptoms by modulating various neural, endocrine, immune, and humoral signaling pathways.

Scientists are trying to develop formulas by studying the relationships between colic and microbiome. Accordingly, if changes in the intestinal microbiota really play a role in infantile colic pathogenesis, it is thought that manipulation of the intestinal microbiome may be a preventive measure and play a therapeutic role in the evolution of these diseases.

Considering that dysbiosis may play a role in infantile colic pathogenesis, there is interest in modulating the gut microbiota, including the use of probiotics for the management of infantile colic. In particular, it is a well-known probiotic that positively modifies the composition of the intestinal microbiota of the Bifidobacterium species and the function of the immune system.

Today, the effect of probiotics added to the diet of the mother and newborn nutrition on the prevention of colic and microbiota content has been evaluated. One study found that when probiotics were added to breast milk, it was effective in reducing the crying time in babies with colic. In studies on the role of probiotics on colic, Lactobacillus species have also been investigated for colic and microbiota, and have been found to reduce crying time in studies showing that they are effective in colic management. When the effects of probiotics given to infants with infantile colic on microbiota are examined, it has been observed in studies that the harmful bacteria types such as H.pylori, Klebsiella, E.coli decrease the amount of beneficial bacteria such as bifidobacterium and lactobacilli. However, studies generally include the addition of probiotics to the diet of babies with colic, and a lack of studies proving that the probiotics given to the mother or foods from natural probiotics (fermented products such as beer, bread, wine, kefir, kumis and cheese) in the mother's diet had a positive effect on the reduction of infantile colic.

This study was planned as a double-blind, randomized placebo-controlled trials in order to evaluate the effect of the probiotic added to the diet of the mothers on infantile colic and the contents of the neonatal intestinal microbiota in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* Mother's ability to speak Turkish,
* Single pregnancy,
* Delivery time is between 37 <GH <42 weeks,
* The mother does not have a chronic disease,
* Vaginal birth,
* The mother's not using antibiotic drugs during pregnancy and postpartum period,
* Neonatal diagnosis of infantile colic,
* Scoring 10 points below the Beck Depression Inventory,
* Smoking of the woman during pregnancy and postpartum period,
* The absence of Intrauterine Growth Retardation (IUGR) or genetic disease in the newborn,
* Birth weight is in the range of 2500-4000 gr.
* No gastrointestinal disease in the newborn,
* 50% of the newborn is feeding on breast milk,
* No more than 24 hours of Early Membrane Rupture (EMR) at birth.

Exclusion Criteria:

* Having problems with the breast in the mother,
* The mother is using probiotics / antibiotics before randomization and during her pregnancy,
* Mothers who are included in the study sample, take part in other clinical studies at the same time.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 31 (Actual)
Dates: Start 2020-10-07 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
crying times | up to 28 days
  reduction of ≥50% of mean daily crying duration. The mothers will provided with a diary(according to the Barr Baby Diary) and they will instructed on how to complete it daily with data concerning administration of daily dose of the study product, number and duration of crying episodes. In addition, mothers will be trained to use stopwatches. They will keep the crying times daily.
microbiota analysis | up to 28 days
  stool sample.

SECONDARY OUTCOMES:
Mother's depression | up to 28 days
  Evaluation of mothers' depression states will be evaluated by filling the "Beck Depression Inventory".
Binding | up to 28 days
  "Maternal Attachment Scale" will be filled in mothers to measure the attachment status between mother and baby.
Babies' height (cm) anthropometric evaluation | up to 28 days
weight (kg) anthropometric evaluation | up to 28 days
head circumference (cm) anthropometric evaluation | up to 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Haseki Eğitim ve Araştırma Hastanesi, Istanbul, Sultangazi, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The study protocol can be shared with other researchers.
Supporting Information: Study Protocol
Time Frame: October 2021- June 2021

REFERENCES:
- [Derived] Yildiz Karaahmet A, Dolgun G, Ozen M, Oguz D. Effect of Maternal Probiotics on Infantile Colic Symptoms and Maternal Quality of Life and Maternal Attachment: A Single-Blind, Randomized Controlled Study. Altern Ther Health Med. 2025 Mar;31(2):18-22. PMID 39715568
- [Derived] Karaahmet AY, Dolgun G, Ozen M. Effects of probiotics on gastrointestinal symptoms, anthropometric measurements, and breastfeeding duration in infants with colic: a randomized control trial. Sao Paulo Med J. 2024 Apr 22;142(4):e2023069. doi: 10.1590/1516-3180.2023.0069.R1.31052023. eCollection 2024. PMID 38655990
- [Derived] Yildiz Karaahmet A, Dolgun G, Ozen M. Probiotics added to maternal nutrition affect infantile colic symptoms and fecal microbiota profile: a single-blind randomized controlled study. Clin Exp Pediatr. 2022 Nov;65(11):547-554. doi: 10.3345/cep.2022.00766. Epub 2022 Sep 23. PMID 36229024